CLINICAL TRIAL: NCT05437393
Title: Children's Adaptive Deep Brain Stimulation for Epilepsy Trial (CADET): Pilot
Acronym: CADET Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); University of Oxford (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 141267
Record Dates: First submitted 2022-06-20; First posted 2022-06-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Lennox-Gastaut Syndrome, Intractable
Keywords: Deep brain stimulation; Neurostimulation; Neuromodulation; Epilepsy; Lennox-Gastaut Syndrome
MeSH Terms: conditions — Epilepsy; Lennox Gastaut Syndrome | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Deep brain stimulation (Experimental): Deep Brain stimulation using a novel device: Bioinduction "Picostim" Deep Brain Stimulation system.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Deep brain stimulation of the centromedian nucleus (bilateral)

SUMMARY:
The CADET Pilot will investigate the safety and feasibility of deep brain stimulation (DBS) to treat children with Lennox-Gastaut syndrome using a novel DBS device (Picostim DyNeuMo-1).

Following a 30-day preoperative/baseline assessment phase, all children will have a neurosurgical procedure to implant the device. Implantation will be followed by a 30-day phase of no stimulation (the device is off / inactive) and then a six-month phase of active stimulation (the device is on / active).

DETAILED DESCRIPTION:
The CADET pilot will be a single-arm, multi-site, interventional clinical trial. This design has been chosen since this is a feasibility and safety trial in a small number of patients and thus does not primarily aim to determine efficacy.

In this pilot clinical trial, four children with drug-resistant LGS will undergo bilateral CMN DBS.

Following the DBS insertion, all children will undergo one month of inactive ('off') DBS in order to allow the lesioning effect of electrode implantation to dissipate. Thereafter, children will receive active ('on') DBS therapy with standard stimulation parameters for six-months. Following the 'on' phase of the trial, the child will then transition into continuing clinical care and will have their stimulation parameters altered according to clinical evaluation.

ELIGIBILITY:
INCLUSION CRITERIA:

Children enrolled in this study must:

1. Be 5-14 years of age at consent.
2. Have a diagnosis of Lennox-Gastaut Syndrome, as determined by:

   * Slow (<3.0Hz) spike-and-wave pattern and/or fast wave pattern (tonic seizures) on EEG for at least six-months months prior to the enrolment into the baseline period
   * History of drop seizures (tonic, atonic, or tonic-clonic) for at least six-months prior to the enrolment into the baseline period
3. Experience at least 10 seizures per month.
4. Have tried and not responded to two or more antiseizure medications prior to enrolment.
5. Be taking one or more anti-seizure medication(s) at a stable dose for at least the four weeks prior and have a parent/guardian(s) who is willing for their child's maintenance anti-seizure drugs to be unaltered for the trial duration.
6. If on a ketogenic diet, have been established on a stable ketogenic diet for at least 12 weeks prior to screening and the parent/guardian(s) to be willing for child to stay on a stable ketogenic for the duration of the trial.
7. Have a parent/guardian(s) who is willing and able to comply with all the requirements of the study, including the completion of the seizure diary and periodic device charging.

   -------------------------------

EXCLUSION CRITERIA:

Children enrolled in this study must not:

1. Have had prior deep brain stimulation insertion.
2. Have an active ('on') vagus nerve stimulator (or active within the six months prior to the baseline period).
3. Have abnormal thalamic anatomy detected on imaging that would render DBS either unsafe or unfeasible.
4. Have a bleeding disorder.
5. Have medical conditions/factors that would increase their anaesthetic risk to an unacceptable level.
6. Have a nickel allergy
7. Be pregnant
8. Participate in contact sports

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Adverse evens | Following 6-months of active stimulation
  Measured according to pre-determined device-related AEs and SAEs, as well as generic AEs and SAEs.
Willingness of the participants/parents/guardians for the participant to be recruited into the study and to undergo the intervention | Following 6-months of active stimulation
  Consent at baseline
Participant completion of the study | Following 6-months of active stimulation
  Completion of all study activities at study exit
Ability of the participant/parent(s)/guardian(s) to re-charge and maintain the device | Following 6-months of active stimulation
  Device recharging is measured using the Picostim event logs

SECONDARY OUTCOMES:
Relative change in parent-reported seizure frequency | Following 6-months of active stimulation (compared to baseline)
  Measured using parent-reported diaries
Relative change in electrographic-recorded seizure frequency | Following 6-months of active stimulation (compared to baseline)
  Measured using serial electroencephalography (EEG)
Relative change in seizure severity | Following 6-months of active stimulation (compared to baseline)
  Measured using the Hague Seizure Severity Scoring questionnaire. Minimum score = 13; maximum score = 52; with higher seizure severity with ascending values.
Relative change in quality of life | Following 6-months of active stimulation (compared to baseline)
  Measured on the Pediatric Quality of Life Inventory (PedsQL) questionnaire. The minimum score is 0 and the maximum score is 100, with improving quality of life with ascending values.
Relative change in quality of life | Following 6-months of active stimulation (compared to baseline)
  Measured on the Impact of Pediatric Epilepsy Scale (IPES) questionnaires. The minimum score is 0 and the maximum score is 100, with improving quality of life with ascending values.

OTHER OUTCOMES:
Radiological correlates of neurophysiological and clinical response to CMN DBS | Following 6-months of active stimulation
  Analysis of pre-trial MRI brain scan in conjunction with relative change in seizure counts measured using parent-reported diaries
Correlates of the scalp EEG with the intracranial recordings (local field potentials) from the DBS device. | Following 6-months of active stimulation
  Analysis of local-field potentials measured from the DBS device in conjunction with data from the encephalography (EEG) data

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No